CLINICAL TRIAL: NCT04834635
Title: The Total Wrapping of the Fundus of the Gastric Excluded Part (FundoRing) Versus Non- Wrapping (Non-banded) Standard Method of Laparoscopic One Anastomosis Gastric Bypass/Mini - Gastric Bypass: A Randomized Controlled Trial
Brief Title: The FundoRingOAGB Versus Non-wrapping (Non-banded) Standard Method of Laparoscopic One Anastomosis Gastric Bypass
Acronym: FundoRingMGB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Society of Bariatric and Metabolic Surgeons of Kazakhstan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FundoRingOAGB
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-01

CONDITIONS: Obesity, Morbid
Keywords: Obesity; Bariatric surgery; One anastomosis gastric bypass; FundoRingOAGB; Fundoplication
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FundoRingOAGB group (Experimental): laparoscopic one anastomosis gastric bypass with the total wrapping of the fundus of gastric excluded part (and suture cruroplasty if present hiatal hernia).
  Interventions: Procedure: FundoRingOAGB
- OAGB group (Active Comparator): laparoscopic one anastomosis gastric bypass (and suture cruroplasty if present hiatal hernia).
  Interventions: Procedure: OAGB

INTERVENTIONS:
Procedure: FundoRingOAGB — laparoscopic one anastomosis gastric bypass with the total wrapping of the fundus of gastric excluded part and with suture cruroplasty if present hiatal hernia
  Arms: FundoRingOAGB group
Procedure: OAGB — laparoscopic one anastomosis gastric bypass with suture cruroplasty if present hiatal hernia
  Arms: OAGB group

SUMMARY:
Currently, one anastomosis gastric bypass (OAGB) or mini-gastric bypass (MGB) is a common bariatric procedure for treating obesity. Weight gain after surgery is a big problem in bariatric practice. Therefore, adjustable bands and rings are used, for example, "FobiRing". But foreign material can cause complications - the erosion of the stomach wall. For this reason, surgeons avoid the use of various mechanical devices on living tissues.

The greatest criticism is of the OAGB for the likelihood of biliary reflux. In case of reflux of bile into the esophagus after surgery, as a rule, a second operation is required with conversion OAGB to the Roux-en-Y method.

In addition, along with obesity, gastroesophageal reflux disease (GERD) are steadily increasing world weight and antireflux surgery must be performed simultaneously with bariatric surgery in obese patients. In these cases, most often in bariatric practice, hiatus cruroraphy is performed, and less often fundoplication using the fundus of the excluded part of the stomach.

We hypothesize that total fundoplication can not only treat GERD but also significant prevent the return of weight like after a banded gastric bypass and prevent postoperative bile reflux in the esophagus.

The aim study is to compare primary outcome as weight loss after total wrapping of the fundus of the gastric excluded part (FundoRing) and non - wrapping (non - banded) standard method of laparoscopic one anastomosis gastric bypass and measure secondary outcome: bile reflux in the esophagus and GERD symptoms.

Methods: Adult participants (n=1000) are randomly allocated to one of two groups:

Experimental surgical bariatric procedure in the first (A) group: patients (n=500) undergo the laparoscopic one anastomosis gastric bypass with the total wrapping of the fundus of gastric excluded part and suture cruroplasty if present hiatal hernia (FundoRingOAGB group); Active comparator surgical bariatric procedure in the second (B) group: patients (n=500) undergo the laparoscopic one anastomosis gastric bypass and with only suture cruroplasty if present hiatal hernia (OAGB group).

DETAILED DESCRIPTION:
One anastomosis Gastric Bypass/Mini Gastric Bypass (OAGB/MGB) is gaining popularity as a primary surgical treatment for morbid obesity.

The aim study is to compare primary outcome as weight loss after total wrapping of the fundus of the gastric excluded part (FundoRing) and non - wrapping (non - banded) standard method of laparoscopic one anastomosis gastric bypass and measure secondary outcome: bile reflux in the esophagus and GERD symptoms.

Methods: Adult participants (n=1000) are randomly allocated to one of two groups:

Experimental surgical bariatric procedure in the first (A) group: patients (n=500) undergo the laparoscopic one anastomosis gastric bypass with the total wrapping of the fundus of gastric excluded part and suture cruroplasty if present hiatal hernia (FundoRingOAGB group); Active comparator surgical bariatric procedure in the second (B) group: patients (n=500) undergo the laparoscopic one anastomosis gastric bypass and with only suture cruroplasty if present hiatal hernia (OAGB group). All patients are then followed up 12, 24, 36 months after surgery where record the changing body mass index and and measure secondary outcome: bile reflux in the esophagus and GERD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* BMI from 30 to 50 kg / m2.
* The person is generally fit for anesthesia (ASA grading 1-2) and surgery.
* The person commits to the need for long-term follow-up.

Exclusion Criteria:

* BMI less than 30 kg / m2 and more than 50 kg / m2.
* Prosthetic (mesh) Hiatal herniorrhaphy or large hiatal hernia;
* Esophageal shortening
* Los Angeles Classification of Oesophagitis (LA grade) C or D reflux esophagitis
* History of surgery on the stomach or esophagus
* Less than 18 or more than 60 years of age
* Not fit for bariatric surgery
* Psychiatric illness
* Patients unwilling or unable to provide informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change of body mass index | Baseline, at 12, 24, 36 months after surgery
  The measure is assessing a change of body mass index. Weight (kg) and height (cm) will be combined with the report of measurement by body mass index (BMI) kg/m2.

SECONDARY OUTCOMES:
Postoperative bile reflux in esophagus | at 12, 24, 36 months after surgery
  The endoscopic finding of postoperative bile reflux in the esophagus
GERD symptoms | Baseline, 12, 24, 36 months after surgery
  Change og GERD symptoms if present GERD or postoperative de Novo GERD symptoms (GERD-HRQL)
Oral glucose tolerance tests | Blood samples for glucose collects at 0, 15, 30, 60, 120, 150 and 180 minutes, while those for insulin collects at 0, 30, 60, 120 and 180 minutes
  A 3-hour oral glucose tolerance tests performs using 75 g glucose
Sigstad score | 6, 12, 24, 36 months after surgery
  Sigstad score for questionnaire of diagnostic the dumping syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Oral Ospanov, Principal Investigator — President of Society of Bariatric and Metabolic Surgeons of Kazakhstan" (SBMSK)
Locations (1):
- Oral Ospanov, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ospanov O, Yeleuov G, Fursov A, Yelembayev B, Fursov R, Sergazin Z, Mustafin A. A laparoscopic one anastomosis gastric bypass with wrapping versus nonwrapping fundus of the excluded part of the stomach to treat obese patients (FundoRingOAGB trial): study protocol for a randomized controlled trial. Trials. 2022 Apr 7;23(1):264. doi: 10.1186/s13063-022-06252-6. PMID 35392958
- [Result] Ospanov O. The Surgical Technique of Primary Modified Fundoplication Using the Excluded Stomach with Simultaneous Gastric Bypass. Obes Surg. 2023 Apr;33(4):1311-1313. doi: 10.1007/s11695-023-06505-6. Epub 2023 Feb 17. PMID 36800158
- [Result] Ospanov O, Yeleuov G, Buchwald JN, Zharov N, Yelembayev B, Sultanov K. A Randomized Controlled Trial of Acid and Bile Reflux Esophagitis Prevention by Modified Fundoplication of the Excluded Stomach in One-Anastomosis Gastric Bypass: 1-Year Results of the FundoRing Trial. Obes Surg. 2023 Jul;33(7):1974-1983. doi: 10.1007/s11695-023-06618-y. Epub 2023 Apr 26. PMID 37099252
- [Derived] Ospanov OB. The Gastric Bypass and Fundoplication in Bariatric Surgery: the Comments on Published Papers and Our Classification of Combination Procedures. Obes Surg. 2021 Oct;31(10):4643-4644. doi: 10.1007/s11695-021-05505-8. Epub 2021 Jun 1. PMID 34059995
- See also: A laparoscopic one anastomosis gastric bypass with wrapping versus nonwrapping fundus of the excluded part of the stomach to treat obese patients (FundoRingOAGB trial): study protocol for a randomized controlled trial — http://pubmed.ncbi.nlm.nih.gov/35392958/
- See also: The Surgical Technique of Primary Modified Fundoplication Using the Excluded Stomach with Simultaneous Gastric Bypass — http://pubmed.ncbi.nlm.nih.gov/36800158/
- See also: A Randomized Controlled Trial of Acid and Bile Reflux Esophagitis Prevention by Modified Fundoplication of the Excluded Stomach in One-Anastomosis Gastric Bypass: 1-Year Results of the FundoRing Trial — https://pubmed.ncbi.nlm.nih.gov/37099252/